CLINICAL TRIAL: NCT03125759
Title: The Association of Omentin and Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xi'an No.3 Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: NDIS001
Record Dates: First submitted 2017-04-01; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Stroke; Brain Ischemia; Adipokines; Mutation
Keywords: Ischemic Stroke; Omentin
MeSH Terms: conditions — Stroke; Brain Ischemia; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood

GROUPS / COHORTS (2):
- Control: patients without any history of stroke
- Ischemic Stroke: patients with an episode of neurological dysfunction caused by focal cerebral, spinal, or retinal infarction within 72 hours.

SUMMARY:
This observational study aims to research whether there is a relationship between omentin and ischemic stroke on the aspects of incidence, severity, and recovery etc.

DETAILED DESCRIPTION:
To study the possible relationship between omentin and ischemic stroke, we intend to recruit the newly found acute ischemic stroke patients and patients without any stroke history and analysis the difference of plasma omentin level and the ITLN, which is the gene symbol of omentin.

ELIGIBILITY:
Inclusion Criteria:

* For ischemic stroke group,acute clinically defined ischemic stroke
* For control group, without any history of stroke

Exclusion Criteria:

For ischemic stroke group

* Hemorrhagic Stroke
* Previous Ischemic Stroke For control group
* The expected life expense less than 3 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: the study population is from primary care clinic, physical examination center, and social volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the odds ratio of omentin plasma concentration between cases and controls | up to 3 years
  The circulation level of omentin will be assessed in cases and controls. Then the odds ratio will be statically analysed to detect whether omentin is asociated with ischemic stroke on protein level.
the frequency difference of single nucleotide polymorphism(SNP) of omentin in the enrolled subjects | up to 3 years
  The SNP will be analysed in the recruited subjects. And the the frequency difference will be calculated to explore if any SNP is related to ischemic stroke.

SECONDARY OUTCOMES:
the NIHSS assessed for functional outcome of stroke | up to 3 years
  NIHSS wil be used to assess neurological status at baseline or the point of stroke, the point of out-patient, 3 month, 6 month, 1 year, 2 year and the 3 year.
the modified Rankin Scale assessed for functional disability | up to 3 years
  Th functional disability will be assessed using the modified Rankin Scale at the time of baseline, out-patient, 3rd month, 6th month, 1st year, 2nd year and the 3rd year after enrollment.
the Barthel index assessed for functional independence in activities | up to 3 years
  The Barthel index at the point of baseline, out-patient, 3rd month, 6th month, 1st year, 2nd year and the 3rd year after enrollment will be assessed for the functional independence in activities.
the number of all cause death | up to 3 years
  The number of all cause of death will be recorded in both groups.
the number of re-stroke in case group | up to 3 years
  Recurrent of stroke will be monitored through out in case group.

CONTACTS AND LOCATIONS:
Overall Officials: Tian Ye, PhD, Principal Investigator — Xi'an No.3 Hospital
Locations (1):
- Xi'an No.3 Hospital, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes